CLINICAL TRIAL: NCT04114513
Title: A Randomized, Placebo-controlled, Double-blinded, Parallel-group, 5-week Study of the Dietary Fibers Intake (Inulin, Pectin, Beta-glucan, Galactooligosaccharides) Influence on the Gut Microbiota Composition and Cardiovascular Risk Factors
Brief Title: Dietary Fibers Effect on the Gut Microbiota Composition
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 lockdown
Sponsor: Atlas Biomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DFI
Record Dates: First submitted 2019-09-27; First posted 2019-10-03 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2019-09

CONDITIONS: Microbiome; Metabolic Syndrome; Cardiovascular Risk Factor; Inflammation; Dyslipidemias
Keywords: Dietary fiber; Gut Microbiota; Cardiovascular risk factors; Lipid metabolism
MeSH Terms: conditions — Metabolic Syndrome; Inflammation; Dyslipidemias | interventions — maltodextrin; Inulin; Pectins; beta-Glucans

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Maltodextrin (Placebo Comparator): Within first 6 days, there will be an increase in the fiber dose: 1st and 2nd days - 2g, 3rd and 4th - 4g per day, 5th and 6th - 6g per day. Starting from the 7th and till the 35th day - 8g per day. Placebo will be given in a powder form to be added to 250 ml of water.
  Interventions: Dietary Supplement: Maltodextrin
- Inulin (Experimental): Within first 6 days, there will be an increase in the fiber dose: 1st and 2nd days - 2g, 3rd and 4th - 4g per day, 5th and 6th - 6g per day. Starting from the 7th and till the 35th day - 8g per day. Placebo will be given in a powder form to be added to 250 ml of water.
  Interventions: Dietary Supplement: Inulin
- Pectin (Experimental): Within first 6 days, there will be an increase in the fiber dose: 1st and 2nd days - 2g, 3rd and 4th - 4g per day, 5th and 6th - 6g per day. Starting from the 7th and till the 35th day - 8g per day. Placebo will be given in a powder form to be added to 250 ml of water.
  Interventions: Dietary Supplement: Pectin
- Beta-glucan (Experimental): Within first 6 days, there will be an increase in the fiber dose: 1st and 2nd days - 2g, 3rd and 4th - 4g per day, 5th and 6th - 6g per day. Starting from the 7th and till the 35th day - 8g per day. Placebo will be given in a powder form to be added to 250 ml of water.
  Interventions: Dietary Supplement: Beta-glucan
- Galactooligosaccharides (Experimental): Within first 6 days, there will be an increase in the fiber dose: 1st and 2nd days - 2g, 3rd and 4th - 4g per day, 5th and 6th - 6g per day. Starting from the 7th and till the 35th day - 8g per day. Placebo will be given in a powder form to be added to 250 ml of water.
  Interventions: Dietary Supplement: Galactooligosaccharides

INTERVENTIONS:
Dietary Supplement: Maltodextrin — NOVAPRODUKT, white powder 5 weeks intervention
  Arms: Maltodextrin
Dietary Supplement: Inulin — BENEO-Orafti, white powder 5 weeks intervention
  Arms: Inulin
Dietary Supplement: Pectin — BANG & BONSOMER GROUP OY, white powder 5 weeks intervention
  Arms: Pectin
Dietary Supplement: Beta-glucan — Tate & Lyle, white powder 5 weeks intervention
  Arms: Beta-glucan
Dietary Supplement: Galactooligosaccharides — FrieslandCampina, white powder 5 weeks intervention
  Arms: Galactooligosaccharides

SUMMARY:
The randomized double-blinded placebo-controlled multicenter study will be held in parallel groups. During 5 weeks the efficacy of different endpoints as a measure of response to the daily intake of dietary fibers (8 g of either inulin, pectin, beta-glucan or galactooligosaccharides) will be evaluated. Gut microbiota composition, lipids levels, inflammation markers, microbiome metabolites, changes in quality of life and stool parameters will be assessed in order to predict individual response in participants without serious chronic diseases

DETAILED DESCRIPTION:
A randomized double-blinded study will include 270 volunteers without clinical manifestations of chronic diseases. Participants will be randomized into one of five arms daily consuming one of the following: placebo (maltodextrin, 8 g), inulin (8 g), pectin (8 g), beta-glucan (8 g) or oligosaccharides (8 g).

The study will include a 5-day screening period and a 5-weeks intervention period.

During screening stage, a volunteer will complete a questionnaire, and the following measurements will be performed: blood levels of glycated hemoglobin, creatinine, lipids, C-reactive protein, anthropometric measurements, as well as cardiovascular risk will be assessed.

Before and after the intervention blood and stool samples will be collected to conduct the following analyses: an extended lipid spectrum analysis, high-sensitivity C-reactive protein, 16S rRNA gut microbiome sequencing, laboratory stool testing, stool fecal short-chain fatty acids analysis. Anthropometric measures, physical examination will be performed for each volunteer. The following questionnaires will be completed: dietary recall questionnaire, SF-36, the Rome Criteria for the Functional gastrointestinal disorders (functional constipation). The assessed scales will include Bristol stool scale, Hospital Anxiety and Depression Scale (HADS), Hamilton Rating Scale for Depression (HRSD).

ELIGIBILITY:
Inclusion Criteria:

* Subject doesn't have any active complaints
* Subject doesn't have any active or acute diseases at the time of enrollment
* Subject signed informed consent

Exclusion Criteria:

* High or very high cardiovascular risk
* Levels of total cholesterol and/or low-density lipoproteins requiring immediate assignment of drug treatment (according to ESC Guidelines for the management of dyslipidaemias, 2019)
* Diabetes mellitus of any type
* HbA1с of 5,7% or higher
* Obesity requiring medical therapy or surgery (according to European Guidelines for Adult Obesity Management, 2019)
* Gastrointestinal diseases in history including ulcerative colitis, Crohn's disease, celiac disease, gallbladder disease (calculous cholecystitis, cholangitis, etc.) not related to functional disorders; liver or pancreas diseases
* Irritable bowel syndrome, abdominal pain of any location and etiology
* Pain syndrome of any localization
* Flatulence
* Oncology diseases
* Mental disorders
* Rheumatoid arthritis or other autoimmune diseases
* Acute infectious diseases or exacerbation of any diseases
* Recent (<3 months) administration of proton pump inhibitors, antimicrobial therapy or surgical intervention
* Recent (<3 weeks) use of probiotics, antacids, nonsteroidal anti-inflammatory drugs, laxatives
* Pregnancy, planning to be pregnant or breast feeding at any point during the study or study enrollment
* Current alcohol/drug abuse (more than 3 points for women and 4 for men according to AUDIT-C questionnaire and/or more than 7 points on the AUDIT questionnaire) or addiction therapy within 12 months prior to screening
* Allergies to any prebiotic or placebo ingredients
* Planned relocation from the home region during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Blood lipids levels | Change from Baseline Blood lipids levels at 5th week
  LDL, HDL, TC, TG, apoB, Lp(a)
Change in Gut microbiota composition | Change from Baseline at 5th week
  Relative abundance of bacterial taxa according to 16S rRNA sequencing data

SECONDARY OUTCOMES:
Change in Fecal short-chain fatty acids | Change from Baseline at 5th week
  Butyrate, propionate and acetate concentrations
Change in High sensitive C-reactive protein | Change from Baseline at 5th week
  Low-grade inflammation assessment
Change in Stool consistency | Change from Baseline at 5th week
  The Bristol stool scale is a diagnostic medical tool designed to classify the form of human faeces into seven categories.
Change in Stool frequency | Change from Baseline at 5th week
  Rome criteria questionnaire. The Rome IV criteria for the diagnosis of irritable bowel syndrome require that patients have had recurrent abdominal pain on average at least 1 day per week during the previous 3 months that is associated with two or more of the following : Related to defecation (may be increased or unchanged by defecation)
Change in Body Composition | Baseline and 5th week
  Bioelectrical impedance analysis
Change in Quality of Life: SF-36 questionnaire | Change from Baseline at 5th week
  According to SF-36 questionnaire The Medical Outcomes Short-Form 36-Item Health Survey (SF-36) It is a self-administered questionnaire comprising 36-items measuring eight dimensions of general HRQOL: physical functioning (10 items), role limitation due to physical health problems (4 items), bodily pain (2 items), general health perceptions (5 items), vitality (4 items), social functioning (2 items), role limitations due to emotional problems (3 items), and general mental health (5 items). In addition to scores for individual dimensions, two summary scores assessing physical and mental dimensions of health and well-being can also be calculated: Physical Component Summary (PCS) score and the Mental Component Summary (MCS) score, respectively
Change in Psychological distress | Change from Baseline at 5th week
  Hospital Anxiety and Depression Scale (HADS) Patients anxiety and depression will be assessed using the HADS : Hospital Anxiety and Depression scale.
  Scores of the HADS scale can be defined as:
  By adding the points of the answers: 1, 3, 5, 7, 9, 11, 13: we obtain the "Total A" which corresponds to the measure of the anxiety, then:
  7 or less: absence of symptomatology; 8 to 10: doubtful symptomatology; 11 and above: certain symptomatology.
  By adding the points of the answers: 2, 4, 6, 8, 10, 12, 14: we obtain the "Total B" which corresponds to the measure of the depression, then:
  7 or less: absence of symptomatology; 8 to 10: doubtful symptomatology; 11 and above: certain symptomatology. The minimal score is 0 and the maximal total score is 42.

CONTACTS AND LOCATIONS:
Locations (1):
- Atlas Medical Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No